CLINICAL TRIAL: NCT04002765
Title: Factors of ILD in Newly Diagnosed Rheumatoid Arthritis
Acronym: FIND-RA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PNEU-ILD-03; 2019/21JUI/269 (Other: CEHF)
Record Dates: First submitted 2019-06-12; First posted 2019-07-01 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Respiratory Function Tests

STUDY DESIGN:
Masking Description: All statistical analysis, including power calculation, will be performed in collaboration with the "Plate-forme en méthodologie statistique" of the UCLouvain. Pre-study estimations revealed that a sample size of 289 patients produces a two-sided 95% confidence interval with a precision (half-width) of 0,04 when the actual proportion is near 0,14.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- New RA patients (Other): * Adults aged 18 to 90 years-old
  * Diagnosis of rheumatoid arthritis (RA) based on ACR-EULAR 2010 criteria
  * Onset of disease duration at least 1 year and at most 10 years prior to inclusion
  Interventions: Diagnostic Test: pulmonary function tests

INTERVENTIONS:
Diagnostic Test: pulmonary function tests — 1. Lung function tests (standard of care)
     1. Dynamic and static volumes (FVC, FEV1, TPC, RV)
     2. Lung diffusion capacity for CO (DLCO)
  2. Chest Xrays
  3. High resolution CT scanner (HRCT)
  Other Names: High-resolution CT scanner

SUMMARY:
To determine factors associated with early RA-ILD (which may be asymptomatic). It is planned to recruit all patients with a newly diagnosed RA (symptoms since less than 3 years). In this study, all relevant demographic and clinical data will be collected. All patients will undergo lung function tests and high-resolution CT-scan of the lungs. Blood sample will be collected for measurement of (1) anti-CCP and rheumatoid factor measurement (good clinical practice) and a specific sample for the detection of the MUC5 promoter variant rs35705950.

Our aim is thus to identify determinants of RA-ILD in the following population:

* Adults aged 18 to 90 years-old
* Diagnosis of rheumatoid arthritis (RA) based on ACR-EULAR 2010 criteria
* Onset of disease duration at least 1 year and at most 10 years prior to inclusion

DETAILED DESCRIPTION:
3. OBJECTIVES The objectives are to (1) detect ILD within a population of early RA and (2) identify potential predictive factors of the development of ILD.

4. METHODS

The study is held in the Rheumatology, Pneumology and Radiology departments of the Cliniques universitaires Saint-Luc and other Belgian hospitals. Patients will be recruited in the rheumatology department (RA consultations). Recruitment will also be possible while patients are hospitalized for a work-up of their RA. At the time of the consultation, the following tests will be performed:

Data collection Clinical data (Standard of Care, SOC)

1. Demographic data
2. Environmental inquiry (smoking status, occupation, domestic exposure)
3. Past medical history
4. Assessment of RA:

   1. ACR/EULAR core set clinical data (joints count, DAS score, HAQ)
   2. Hand and feet Xrays Biological assessment

<!-- -->

1. Biological data (SOC)

   1. CRP
   2. Rheumatoid factor
   3. Anti-CCP antibodies
   4. Antinuclear antibodies
2. Genetic sampling (non-SOC) a. Detection of the rs35705950 variant for MUC5B promoter Lung assessment (SOC)

1. Lung function tests (standard of care)

1. Dynamic and static volumes (FVC, FEV1, TPC, RV)
2. Lung diffusion capacity for CO (DLCO) 2. Chest Xrays 3. High resolution CT scanner (HRCT)

<!-- -->

1. Good clinical practice (INAMI/RIZIV)
2. Including expiratory slices (detection of early air trapping) Primary outcome Detection of an interstitial lung disease associated with RA. RA-ILD is defined by the presence of reticulations, ground-glass opacity and/or honeycombing at HRCT not explained by another cause (i.e. cardiac disease, infection or neoplasia). The expected frequency of RA-ILD is 14% (based on local retrospective study on 1000 RA patients).

   Secondary outcomes 1. Proportion of different ILD subtypes (usual interstitial pneumonia, non-specific interstitial pneumonia, others) 2. Detection of non-ILD lung involvement of RA including:

   - Rheumatoid nodules

   - Emphysema

   - Bronchiectasis not related to an ILD

   - Bronchiolitis obliterans 3. Proportion of patients carrying the variant rs35705950 of the MUC5B promoter 4. Proportion of patients with anti-CCP antibodies 5. Proportion of patients with a relevant toxic exposure (smoking, drug, occupational or domestic exposure) 4.4 Expected timeline

   Start of recruitment: 01-July-2019 End of recruitment: 31-Dec-2022 Based on our local recruitment of RA patients, it is expect to recruit 300 patients.

   4.5. Méthodes d'analyse des données y compris des données manquantes, inutilisées ou Erronées All statistical analysis, including power calculation, will be performed in collaboration with the "Plate-forme en méthodologie statistique" of the UCLouvain. Pre-study estimations revealed that a sample size of 289 patients produces a two-sided 95% confidence interval with a precision (half-width) of 0,04 when the actual proportion is near 0,14.

   5. POPULATION 5.1 Inclusion criteria

   - Adults aged 18 to 90 years-old

   - Diagnosis of rheumatoid arthritis (RA) based on ACR-EULAR 2010 criteria

   - Onset of disease duration at least 1 year and at most 10 years prior to inclusion 5.3 Exclusion criteria

   - Pregnancy
   * Inability to provide informed consent
   * Inability to perform lung function tests or to comply with the protocol
   * Active pulmonary infection 6. CONFIDENTIALITY We will ensure study data confidentiality and anonymization (Law of 08 December 1992 on Privacy Protection, Law of 22 August 2002 on patients' rights and GDPR): A number will identify each subject. Only the PI and co-PI will have the ability to link the subject's number to his/her medical file. All data will be stored in a database, which will be held on CUSL' computer server. Access to data will be secured by (1) identification of PI and co-PI on their office desk and (2) by a specific password.

     7. ETHICS This protocol is submitted for approval to our local Ethics committee (Comité d'Ethique Hospitalo-facultaire CUSL-UCLouvain).

     8. INSURANCE

   An appropriate insurance will be taken to cover the risks ("assurance sans faute").

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 90 years-old
* Diagnosis of rheumatoid arthritis (RA) based on ACR-EULAR 2010 criteria
* Onset of disease duration at least 1 year and at most 10 years prior to inclusion

Exclusion Criteria:

* Pregnancy
* Inability to provide informed consent
* Inability to perform lung function tests or to comply with the protocol
* Active pulmonary infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence of an interstitial lung disease | from enrollment of patient to 3 months post enrollment
  Detection of an interstitial lung disease associated with RA. We define RA-ILD by the presence of reticulations, ground-glass opacity and/or honeycombing at HRCT not explained by another cause (i.e. cardiac disease, infection or neoplasia).

SECONDARY OUTCOMES:
Proportion of different ILD subtypes | from enrollment of patient to 3 months post enrollment
  usual interstitial pneumonia, non-specific interstitial pneumonia, others
Proportion of patients presenting with a non-ILD lung involvement of RA | from enrollment of patient to 3 months post enrollment
  Non-ILD lung involvement is a composite of the following variables: rheumatoid nodules, emphysema, bronchiectasis and bronchiolitis obliterans
rs35705950 variant of the MUC5B promoter | from enrollment of patient to 3 months post enrollment
  Proportion of patients carrying the variant rs35705950 of the MUC5B promoter
anti-CCP antibodies | from enrollment of patient to 3 months post enrollment
  Proportion of patients with anti-CCP antibodies
relevant exposure | from enrollment of patient to 3 months post enrollment
  Proportion of patients with a relevant toxic exposure (smoking, drug, occupational or domestic exposure)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Froidure, MD PhD, Study Director — Cliniques universitaires Saint-Luc- Université Catholique de Louvain; Patrick Durez, MD PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain; Benoît Ghaye, MD PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (2):
- Belgium (2):
  - Cliniques universitaires Saint-Luc, Brussels
  - CHU-UCL Namur - Site Mont-Godinne, Yvoir

IPD SHARING:
Plan to Share IPD: No
We will ensure study data confidentiality and anonymization (Law of 08 December 1992 on Privacy Protection, Law of 22 August 2002 on patients' rights and GDPR): A number will identify each subject. Only the PI and co-PI will have the ability to link the subject's number to his/her medical file. All data will be stored in a database, which will be held on CUSL' computer server. Access to data will be secured by (1) identification of PI and co-PI on their office desk and (2) by a specific password.